CLINICAL TRIAL: NCT01370941
Title: The Effect of Chymosin on the Intestinal Absorption of Calcium: A Randomized Controlled Cross-over Trial
Brief Title: The Effect of Chymosin on the Intestinal Absorption of Calcium
Acronym: Chymosin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Chymo-01; 20110007 (Registry Identifier: The ethical Committees Region Mid-Jytland)
Record Dates: First submitted 2011-04-27; First posted 2011-06-10 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Osteoporosis; Osteopenia
Keywords: Chymosin; 24H urine calcium excretion; Calcium absorption; Intestinal Absorption of Calcium
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug A: Chymosin (Active Comparator): A: 5 drops of Chymosin is added to ½ a liter of milk. This is to be consumed during breakfast.
  Interventions: Dietary Supplement: Drug A Chymosin
- Drug B: Placebo (Placebo Comparator): B: 5 drops of placebo (water) is added to ½ a liter of milk. This is to be consumed during breakfast.
  Interventions: Dietary Supplement: Drug B: Placebo

INTERVENTIONS:
Dietary Supplement: Drug A Chymosin — Five drops of chymosin is added to ½ a liter of milk. This is to be consumed during breakfast.
  Other Names: Chy-max plus IMCU200
  Arms: Drug A: Chymosin
Dietary Supplement: Drug B: Placebo — B: Five drops of placebo (water) is added to ½ a liter of milk. This is to be consumed during breakfast.
  Other Names: Water
  Arms: Drug B: Placebo

SUMMARY:
An adequate calcium intake is important for bone turnover and the risk of developing osteoporosis. Yet many studies have documented that supplementation with calcium tablets are often associated with a poor compliance, therefore it is important to explore ways to better calcium influx.

Calcium consumed through dairy products must first be cleaved from the molecules which it is bound to before it can be absorbed. Chymosin is an enzyme which cleaves the protein binding between some amino acids in κ-casein. The reaction occurs after ingestion of milk and causes a process whereby the time the milk is staying gastrointestinal tract is extended, this can lead to enhanced uptake of calcium.

When the body's calcium balance is in equilibrium excretion in urine (24 h) in roughly the size of the intake, whereby a measurement of circadian urine excretion of calcium can determine the amount of calcium absorbed from the intestine.

The investigators want to clarify whether the addition of chymosin to milk increases calcium absorption. Secondary to explore issues of significance for this effect, including vitamin D status and amount of daily calcium intake and whether a change in calcium absorption has immediate effects on bone turnover (measured as plasma osteocalcin, bone specific alkaline phosphatase (BSAP), and the renal excretion of cross-linked N-terminal telopeptide of type 1 collagen (NTx/Cr) ratio) and on the parathyroid function (measured as PTH). Finally we will explore relations between bone mineral density (BMD) and the measured parameters (in terms of P-PTH, P-25OHD, P-1,25(OH)2D, P-osteocalcin, P-BSAP, and U-NTx/Cr).

DETAILED DESCRIPTION:
Background:

Osteoporosis is a frequent disease. Allegedly, more than 500,000 Danes are diagnosed with osteoporosis and, in consequence, seems every year more than 20,000 fractures. A number of factors are known to increase the risk of osteoporosis, including a low daily intake of calcium.

Several clinical trials with calcium supplements for adults (with or without simultaneous supplementation of vitamin D) have shown an increase in bone mineral density (Bone Mineral Density, BMD) and reduction the risk of fractures. Similarly, several studies have shown that high milk intake during childhood and adolescence may increase bone mass and reduce the risk of fractures later in life.

Since an adequate calcium intake is important for bone turnover and the risk of developing osteoporosis, it is important to explore ways to better calcium influx. Several studies have documented that supplementation with calcium tablets are often associated with a poor compliance - people do not remember to take the tablets. It is therefore desirable to find methods that can increase the intake of the amount of calcium which occurs naturally in the diet.

Calcium consumed through dairy products must first be cleaved from the molecules which it is bound to before it can be absorbed. Various methods have been tried to optimizing the amount of calcium absorbed from dairy products, including the addition of so called fructo-oligosaccharides (FOSS) and casein phosphopeptides (CPPs).

Chymosin is an enzyme which cleaves the protein binding between some amino acids in κ-casein. The reaction occurs after ingestion of milk and causes a process whereby the time the milk is staying gastrointestinal tract is extended, this can lead to enhanced uptake of calcium. When the body's calcium balance is in balance the excretion in urine (24 h)is in roughly the size as the intake. Therefore a measurement of circadian urine excretion of calcium can determine the amount of calcium absorbed from the intestine.

Purpose and hypothesis:

Primarily the study intends to clarify whether the addition of chymosin to milk increases the intestinal calcium absorption. Secondary to explore issues of significance for this effect, including vitamin D status and amount of daily calcium intake, and whether a change in calcium absorption has immediate effects on bone turnover (measured as plasma osteocalcin, plasma bone specific alkaline phosphatase, and the renal excretion of cross-linked N-terminal telopeptide of type 1 collagen (NTx/Cr) ratio) and on the parathyroid function (measured as PTH). Finally we will explore relations between bone mineral density (BMD) and the measured parameters (in terms of P-PTH, P-25OHD, P-1,25(OH)2D, P-osteocalcin, P-BSAP, and U-NTx/Cr).

Design:

The study is conducted as a randomized double-blinded controlled cross-over trial in which 125 healthy subjects will be asked to drink a glass of milk with or without added chymosin at two occasions. The two time two test days will be separated by 10-18 days. Neither study participants nor the staff conducting the investigation (investigator) will while the trial will be conducted know on which day of the trial which milk contains chymosin (double-blinded). About chymosin added to milk on the first or second test day will be determined by lot (randomized study).

Study Population:

Healthy participants in the agegroup of 25-40 years old are recruited. From the central personal register (CPR register) a list of young people living in the Aarhus area is drawn up, followed by sending out a direct letter asking for participation in the study. At the same time a questionnaire will clarify whether participation is possible, i.e. whether the criteria for participation in the survey are meet.

ELIGIBILITY:
Inclusion Criteria:

* A stable daily intake of calcium on estimated 500-1200 mg, of which dairy products are minimum 500 mg
* Speak and read Danish.
* Written consent after verbal and written information

Exclusion Criteria:

* Known lactose intolerance / milk allergy
* Use of calcium supplements in tablet or powder
* Intake of vitamin D supplements exceeding 10 micro grams/day
* A habitual dietary calcium intake exceeding 1200 mg/day
* Impaired renal function (plasma creatinine >150 micro mol/L)
* Impaired liver function (plasma ALT >200 U/L, alkaline phosphatase >400 U/L).
* Previous or present malignancies(including metastases).
* sarcoidosis or second granulomatous disease which has caused hypercalcaemia
* Pregnancy, breastfeeding
* Postmenopausal women
* Disease or treatment with drugs known to affect calcium homeostasis, including diuretics, osteoporosis agents, lithium, steroids, etc..
* Pledged due to chronic alcoholism.
* Severe medical or social problems which makes it unlikely that the participant can complete the survey
* Lack of willingness / desire to participate

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The effect of the intervention on the 24 hours urine excretion of calcium corrected for creatinine | Two time two days over an eighteen days period
  The effect of the intervention on the 24 hours urine excretion of calcium corrected for creatinine

SECONDARY OUTCOMES:
The effect of plasma 25-hydroxyvitamin D and 1,25-dihydroxyvitamin D levels on the amount of calcium absorbed and the potential impact of chymosin | Two time two days over an eighteen days period
  Vitamin D: The importance of plasma 25-hydroxyvitamin D and 1,25-dihydroxyvitamin D on the amount of calcium absorbed and the potential impact of chymosin.
The immediate biological effects of the intervention on P-PTH, and bone turnover (P-osteocalcin, P-BSAP, U-NTX) | Two time two days over an eighteen days period
  The immediate biological effects of the intervention on parathyroid function (PTH) and bone turnover (P-osteocalcin, plasma bone specific alkaline phosphatase, and the renal excretion of cross-linked N-terminal telopeptide of type 1 collagen (NTx/Cr) ratio).
Relations between bone mineral density (BMD) and the measured parameters (P-25OHD, P-1,25(OH)2D), P-PTH, P-osteocalcin, P-BSAP, U-NTx/Cr) | Will be measured one time at one of the two time two days over an eighteen days period
  To explore relations between bone mineral density (BMD) and the measured parameters (P-25OHD, P-1,25(OH)2D), P-PTH, P-osteocalcin, P-BSAP, U-NTx/Cr).

CONTACTS AND LOCATIONS:
Overall Officials: Leif Mosekilde, Professor, Principal Investigator — Aarhus University Hospital, THG
Locations (1):
- Ward 900, Osteporosis clinic, Aarhus University Hospital, THG, Aarhus, Jutland, Denmark

REFERENCES:
- [Derived] Moller UK, Jensen LT, Mosekilde L, Rejnmark L. Effects of adding chymosin to milk on calcium homeostasis: a randomized, double-blind, cross-over study. Calcif Tissue Int. 2015 Feb;96(2):105-12. doi: 10.1007/s00223-014-9942-8. Epub 2014 Dec 18. PMID 25515208